CLINICAL TRIAL: NCT00351728
Title: Combined PET/CT Imaging for the Early Detection of Ocular Melanoma Metastasis Compared to CT Scanning Alone
Status: Completed | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UCLA IRB #05-04-016
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Ocular Melanoma; Choroidal Melanoma; Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Patients diagnosed with ocular melanoma consent to participate in the study. Combined PET/CT scans of the whole body are performed at baseline, three months later, and six months after that for a total of three combined scans in the first year. Subsequently, these combined scans will be performed at 6-monthly intervals for a total of two combined scans per year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of ocular melanoma (a pigmented malignant tumor) involving the choroid and/or ciliary body (the blood vessel layer in the back of the eye and/or the part of the eye behind the iris).
2. Patients 18 years of age or older.
3. Patients able to give informed consent.

Exclusion Criteria:

1. Patients who refuse to participate in the study.
2. Patients who are unable to cooperate with or cannot undergo PET/CT scanning.
3. Patients who will be moving out of the area of UCLA during the ten years of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: choroidal melanoma patients
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2006-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara A McCannel, MD, PhD, Principal Investigator — Jules Stein Eye Institute, UCLA
Locations (1):
- Jules Stein Eye Institute, Los Angeles, California, United States